CLINICAL TRIAL: NCT02814448
Title: CryoPen: An Innovative Treatment for Cervical Precancer in Low-Resource Settings
Brief Title: An Innovative Treatment for Cervical Pre Cancer
Acronym: CryoPen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Basic Health International (Other); CryoPen, Inc. (Other); University of Southern California (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-296; UH2CA189883 (NIH)
Record Dates: First submitted 2016-06-13; First posted 2016-06-27 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CO2 standard cryotherapy- double freeze (Active Comparator): Double freeze treatment consists of three-minute freeze, five-minute thaw, three-minute freeze
  Interventions: Device: CO2 standard cryotherapy
- CO2 standard cryotherapy- single freeze (Active Comparator): Single freeze treatment consists of one five-minute freeze
  Interventions: Device: CO2 standard cryotherapy
- CryoPen- double freeze (Active Comparator): Double freeze treatment consists of three-minute freeze, five-minute thaw, three-minute freeze
  Interventions: Device: CryoPen
- CryoPen- single freeze (Active Comparator): Single freeze treatment consists of one five-minute freeze
  Interventions: Device: CryoPen
- Thermocoagulator (Experimental): Single heat application at 100 ºC for 40 seconds
  Interventions: Device: Thermocoagulator

INTERVENTIONS:
Device: CryoPen — Provides a means of freezing tissue without the use of gases or liquids
  Arms: CryoPen- double freeze; CryoPen- single freeze
Device: CO2 standard cryotherapy — Standard therapy using carbon dioxide for freezing of tissue
  Arms: CO2 standard cryotherapy- double freeze; CO2 standard cryotherapy- single freeze
Device: Thermocoagulator — The use of heat produced by high-frequency electric current to bring about local destruction of tissues
  Arms: Thermocoagulator

SUMMARY:
The purpose of this study is to test two innovative devices, the CryoPen® and thermocoagulator, against gas-based cryotherapy to determine whether the novel devices produce equivalent or improved destruction of cervical tissue compared to gas-based cryotherapy. Tissue destruction with single freeze versus double freeze treatments with the CryoPen and gas-based cryotherapy will also be compared.

DETAILED DESCRIPTION:
The primary objectives of the study are to test the hypothesis that the CryoPen® and thermocoagulator provide a non-inferior depth of cervical tissue necrosis compared with traditional CO2-based cryotherapy and to test single versus double freeze applications. The secondary objectives of the study are to determine if the CryoPen® or thermocoagulator achieves a depth of necrosis of 3.5 mm, the accepted depth required for eradicating 95% of cervical precancer, and to observe the relationship between depth of necrosis and variations in cervical anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 and 65 years old.
* Scheduled for a hysterectomy for reasons other than cervical precancer or cancer
* Diagnosis of uterine, endometrial, ovarian or other cancer that does not jeopardize the tissue of the cervix is permitted
* Histological evaluation of the cervix does not interfere with the woman's current diagnosis
* Woman consents to participate after being informed about the study
* Normal Pap Smear or HPV test in the past 3 years

Exclusion Criteria:

* Pregnancy
* History of cervical surgery in past 5 years
* Presence of cervical lesion pre-invasive or invasive on the cervix *
* Current Pelvic Inflammatory Disorder or severe acute cervicitis
* Cervix shape disfigured or hard to reach

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Cremer, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- Hospital 1 de Mayo del Instituto Salvadoreño del Seguro Social, San Salvador, El Salvador
- Instituto Nacional de Enfermedades Neoplásicas, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were between the ages of 25 and 65 to be eligible for the study
Period: Overall Study
Arm/Group | CO2 Standard Cryotherapy- Double Freeze | CO2 Standard Cryotherapy- Single Freeze | CryoPen- Double Freeze | CryoPen- Single Freeze | Thermocoagulator
Started | 27 | 24 | 26 | 25 | 28
Completed | 27 | 24 | 25 | 25 | 26
Not Completed | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO2 Standard Cryotherapy- Double Freeze | CO2 Standard Cryotherapy- Single Freeze | CryoPen- Double Freeze | CryoPen- Single Freeze | Thermocoagulator | Total
Number analyzed (Participants) | 27 | 24 | 26 | 25 | 28 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 26 | 25 | 28 | 130
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.46 (6.44) | 45.5 (6.53) | 45.92 (5.82) | 44.65 (5.91) | 45.35 (6.05) | 45.37 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 26 | 25 | 28 | 130
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  El Salvador | 15 | 15 | 16 | 15 | 18 | 79
  Peru | 12 | 9 | 10 | 10 | 10 | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Depth of Necrosis Achieved With the LMIC-adapted CryoPen and the Thermocoagulator Compared to Mean Depth of Necrosis Achieved With CO2-based Cryotherapy
Time Frame: 24-48 hours after treatment
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | CO2 Standard Cryotherapy- Double Freeze | CO2 Standard Cryotherapy- Single Freeze | CryoPen- Double Freeze | CryoPen- Single Freeze | Thermocoagulator
Number analyzed (Participants) | 27 | 24 | 25 | 25 | 26
millimeters | 6.0 (1.6) | 5.6 (1.9) | 5.3 (1.2) | 5.5 (1.3) | 3.5 (0.9)

2. Secondary Outcome: Mean Pain During Treatment Reported by Patients Treated With Double and Single Freeze CO2 Cryotherapy, Double and Single Freeze CryoPen and Thermoablation
Description: Scale Title: Pain scale during treatment Minimal value = 0 (no pain) Maximum value = 10 (most pain) This is a one item 11-point scale to measure self-reported pain during each of the treatments which lasted between 40 seconds (thermoablation) and 13 minutes (double freeze cryotherapy and double freeze CryoPen).
Time Frame: 40 seconds to 13 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CO2 Standard Cryotherapy- Double Freeze | CO2 Standard Cryotherapy- Single Freeze | CryoPen- Double Freeze | CryoPen- Single Freeze | Thermocoagulator
Number analyzed (Participants) | 27 | 24 | 25 | 25 | 26
units on a scale | 2.2 (1.0) | 1.8 (0.8) | 2.5 (1.4) | 2.6 (1.4) | 4.1 (2.3)

ADVERSE EVENTS:
Arm/Group | CO2 Standard Cryotherapy- Double Freeze | CO2 Standard Cryotherapy- Single Freeze | CryoPen- Double Freeze | CryoPen- Single Freeze | Thermocoagulator
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24 | 0/26 | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/26 | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/26 | 0/25 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes